CLINICAL TRIAL: NCT06437041
Title: Effect of Antibiotic Pretreatment on the Efficacy of WMT in the Treatment of Irritable Bowel Syndrome in Adults: a Multi-center, Randomized, Placebo-controlledClinical Study
Brief Title: Effect of Antibiotic Pretreatment on the Efficacy of WMT in the Treatment of Irritable Bowel Syndrome
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faming Zhang (Other)
Responsible Party: Sponsor-Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Organization: The Second Hospital of Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WMT-ABx-IBS-202405
Record Dates: First submitted 2024-05-24; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Irritable Bowel Syndrome
Keywords: Irritable bowel syndrome; washed microbiota transplantation; antibiotic pretreatment; randomized controlled trial; transendoscopic enteral tube
MeSH Terms: conditions — Irritable Bowel Syndrome | interventions — Ornidazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Patients will receive three enemas of ornidazole 0.5g+50ml saline through the TET tube, followed by WMT once daily for a duration of 3 days.
  Interventions: Drug: Ornidazole
- Control (Placebo Comparator): Patients will receive three enemas of a placebo of equal volume through the TET tube, followed by WMT once daily for a duration of 3 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ornidazole — Patients will receive three consecutive enemas of ornidazole 0.5g+50ml saline through the TET tube, followed by WMT treatment once daily for a duration of 3 days.
  Other Names: washed microbiota transplantation
  Arms: Treatment
Drug: Placebo — Patients will receive three consecutive enemas of placebo of equal volume through the TET tube, followed by WMT treatment once daily for a duration of 3 days
  Other Names: washed microbiota transplantation
  Arms: Control

SUMMARY:
This is a randomized controlled trial to explore the efficacy of antibiotic pretreatment on the efficacy of WMT in the treatment of Irritable bowel syndrome in adults: a multi-center, randomized, placebo-controlled clinical study

DETAILED DESCRIPTION:
All included in the standard but do not accord with standard of any rule out subjects will be included in this study. Demographic characteristics, Gastrointestinal Symptoms Rating Scales（GSRS），IBS Symptom Severity Scaleand(IBS-SSS) 、Pittsburgh Sleep Quality Index（PSQI）、Self-rating Anxiety Scale（SAS）、Self-rating Depression Scale（SDS）and clinical outcomes will be collected. After the treatment, the efficacy and safety will be evaluated during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed the informed consent, age 18 years old or more, men and women all can;
2. According to the Roman IV standard diagnosis of IBS: recurrent abdominal pain or discomfort, weekly attacks within the past 3 months at least 3 d, accompanied by the following two and two or more:

(1) associated with defecation; (2) changes in defecation frequency; (3) changes in stool characteristics (appearance).

The following symptoms were not included in the diagnostic criteria but supported the diagnosis: (1) abnormal bowel frequency: bowel movements less than 3 times per week or more than 3 times per day; (2) the excrement characters and abnormal: dry bulb dung or hard dung, or paste dung/dilute waste water; (3) bowel effort; (4) Defecation urgency, endless defecation, mucus excretion and abdominal distension.

Diagnostic considerations: (1) Diagnosis should be based on the exclusion of organic diseases; (2) the intestinal symptoms of irritable bowel syndrome has certain characteristics, such as abdominal pain or discomfort with bowel movements, this group of symptoms is different from the other functional bowel disease, such as functional constipation, functional diarrhea, functional abdominal pain). (3) Irritable bowel syndrome often coexists with other functional gastrointestinal disorders.

3. The subjects or their legal representatives gave informed consent, fully understood the purpose of the study, were able to communicate well with the researchers, and understood and complied with the requirements of the study.

Exclusion Criteria:

* Subjects meeting any of the following exclusion criteria must be excluded from the study:

  1. The patient was accompanied by other mental disorders besides anxiety and depression.
  2. Combined with the results of colonoscopy within the past 24 months, the patient has an organic lesion of the digestive tract (e.g., tumor, inflammation, anal fissure, Crohn's disease, ulcerative colitis, intestinal adhesion, intestinal tuberculosis, etc.).
  3. Has a history of major surgery within 3 months or a history of severetrauma, and recovery is not completely;

  6. There are contraindications to colonic transendoscopic intestinal tubeimplantation, such as severe intestinal stenosis, obstruction, deep ulcer,and high risk of operation perforation; Severe ulcers or a large numberof pseudopolyps exist in the fixed area of titanium clips, which are notsuitable for fixation. The subjects' behavior was seriously uncontrolled.

  7. Any of the following abnormalities in cardiac function and performance:a. According to the New York Heart Association (NYHA) cardiacfunction classification, cardiac function grade # or above;b. new onset myocardial infarction or unstable angina pectoriswithin 6 months;c. ECG showed QTc prolongation (QTc≥ 450ms in men and≥470ms in women);d. Drug-refractory atrial arrhythmias and drug-refractory ventriculararrhythmias (including grade 2 or higher atrioventricular block).

  8. Patients with poor lung function that is considered by the investigatorto have an impact on the study treatment, such as patients with acuteexacerbation of COPD or patients requiring long-term use of oral orintravenous steroids for control (except inhalers/sprays); 9. No control autoimmune disease and/or need long-term use of hormone(except local external use sex); 10. Patients with metabolic diseases and poorly controlled by drugs(such as thyroid dysfunction), or patients with metabolic diseases accompanied by gastrointestinal function complications (such as gastrointestinal autonomic nerve dysfunction, diabetic gastroparesis,etc.) 11. Suffering from reproductive system diseases (including but not limited toovarian cysts, endometriosis, primary dysmenorrhea, etc.) that may lead to abdominal pain; 12. Significant laboratory abnormalities that, in the judgment of theinvestigator, may affect the safety of the subjects or the completion ofthe clinical study, including:A) the hemoglobin < 100 g/L; B) Serum creatinine ≥1.5 times theupper limit of normal (ULN) C) abnormal liver function, defined asAST>1.5×ULN and/or ALT>1.5×ULN and/or total bilirubin >1.5×ULN;D) blood clotting function: PLT acuities were 80 x 109 / L, APTT > 1.5 xULN, PT > 1.5 x ULN, INR > 1.5 x ULN; E) abnormal results or defecateoccult blood stool and has prompted the clinical significance of thegastrointestinal tract.

  13. Have active hepatitis (requiring or taking long-term treatment), HIV, oractive tuberculosis; 14. A history of drug or alcohol abuse (i.e., drinking more than 14 servings per week of beer, 45 mL of 40% spirits, or 150 mL of wine) or substance abuse; 15. The known allergic to research similar drugs, drugs or accessories; 16. Use of anti-infective drugs (antibiotics, antifungal, antiviral) within 14days before enrollment, or need anti-infective treatment at enrollmentevaluation; 17. Drugs and supplements that affect gastrointestinal motility and functioncannot be stopped during the study, including but not limited to:antibiotics such as erythromycin; Drugs that modulate the intestinal microecology, such as probiotics such as Bifidobacterium; Theparasympathetic nerve inhibitors, some scopolamine and atropine,belladonna, etc; Muscle relaxants, such as succinylcholine; Opioid preparations; Drugs thatinhibit gastric acid secretion; 18. Pregnant or lactating women, or refusing to use an effectivecontraceptive method within 3 months after the last dose of treatment; 19. 3 months prior to dosing involved in drug interventional clinical trials; 20. Suffering from malignant tumors;21. There were other circumstances that the investigator consideredinappropriate for participatin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
Gastrointestinal Symptoms Rating Scales（GSRS） | One-week, Four-week and Eight-week post-WMT
  Gastrointestinal Symptom Rating Scale (GSRS) included 5 items: abdominal pain (3 items), reflux (2 items), dyspepsia (4 items), diarrhea (3 items) and constipation (3 items). The severity of each symptom was assessed using a 4-point Likert scale, with a score of 0 indicating no symptoms and a score of 3 indicating very severe symptoms.
IBS Symptom Severity Scaleand(IBS-SSS) | One-week, Four-week and Eight-week post-WMT
  IBS symptom severity scale (IBS-SSS) consists of five items, which assess the severity of abdominal pain, the frequency of abdominal pain, the degree of abdominal distention and discomfort, the satisfaction of bowel habit and behavior, and the impact of intestinal symptoms on life. Each item was divided into 5 levels, increasing by 20 points, and the total score was 500 points. A score of 75 to 175 is mild, 176 to 300 is moderate, and more than 300 is severe.

SECONDARY OUTCOMES:
Pittsburgh Sleep Quality Index（PSQI） | One-week, Four-week and Eight-week post-WMT
  PSQI was used to assess the sleep quality of the subjects in the last month. It consisted of 19 self-rated items and 5 patient-rated items.
Self-rating Anxiety Scale（SAS） | One-week, Four-week and Eight-week post-WMT
  Self-rating anxiety Scale (SAS) is a self-rating scale used to evaluate the subjective feelings of patients with anxiety. It contains 20 items and is divided into 4 grades.
Self-rating Depression Scale（SDS） | One-week, Four-week and Eight-week post-WMT
  Self-rating Depression Scale,SDS is a self-rating scale that measures subjective feelings of depression. It contains 20 items and is scored on a 4-point scale.

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh P, Alm EJ, Kelley JM, Cheng V, Smith M, Kassam Z, Nee J, Iturrino J, Lembo A. Effect of antibiotic pretreatment on bacterial engraftment after Fecal Microbiota Transplant (FMT) in IBS-D. Gut Microbes. 2022 Jan-Dec;14(1):2020067. doi: 10.1080/19490976.2021.2020067. PMID 35014601
- [Background] Xu J, Xu H, Guo X, Zhao H, Wang J, Li J, He J, Huang H, Huang C, Zhao C, Li Y, Zhou Y, Peng Y, Nie Y. Pretreatment with an antibiotics cocktail enhances the protective effect of probiotics by regulating SCFA metabolism and Th1/Th2/Th17 cell immune responses. BMC Microbiol. 2024 Mar 18;24(1):91. doi: 10.1186/s12866-024-03251-2. PMID 38500062
- [Background] Keshteli AH, Millan B, Madsen KL. Pretreatment with antibiotics may enhance the efficacy of fecal microbiota transplantation in ulcerative colitis: a meta-analysis. Mucosal Immunol. 2017 Mar;10(2):565-566. doi: 10.1038/mi.2016.123. Epub 2016 Dec 21. No abstract available. PMID 28000680